CLINICAL TRIAL: NCT01626612
Title: De-escalation of Empirical Antimicrobial Therapy Study in Severe Sepsis: A Randomized Clinical Trial (DEA Study)
Brief Title: De-escalation of Empirical Antimicrobial Therapy Study in Severe Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002297-22; 2011 -10 (Other: AP HM)
Record Dates: First submitted 2012-06-04; First posted 2012-06-25 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- a strategy based on de-escalation (Experimental)
  Interventions: Procedure: streamlining of the empirical antimicrobial therapy
- a conservative strategy (Active Comparator)
  Interventions: Procedure: continuation of the empirical antimicrobial therapy

INTERVENTIONS:
Procedure: continuation of the empirical antimicrobial therapy — ALL THE ANTIBACTERIAL IN WORN SYSTEMATIC
  Arms: a conservative strategy
Procedure: streamlining of the empirical antimicrobial therapy — ALL THE ANTIBACTERIAL IN WORN SYSTEMATIC
  Arms: a strategy based on de-escalation

SUMMARY:
Rational: Severe sepsis is one of the leading cause of mortality in intensive care unit patients. Early initiation of an appropriate empirical antimicrobial therapy is associated with improved outcomes. In order to avoid an increase of selection pressure and the emergence of multidrug resistant pathogens, guidelines recommend to streamline the antimicrobial therapy after the identification of the pathogen responsible for infection. This strategy has been evaluated in several observational studies. However, at the bedside, few randomized clinical trials tested this strategy prospectively.

Method: the investigators conduct a randomized clinical trial comparing a strategy based on de-escalation (streamlining of the empirical antimicrobial therapy) and a conservative strategy (continuation of the empirical antimicrobial therapy). The investigators first aim was to show that a strategy based on de-escalation is not inferior to a conservative strategy in terms of intensive care unit length of stay. Secondary aims are to compare the rate of mortality rate, the emergence of multidrug resistant pathogens, and the feasibility of de-escalation. The study is performed in nine intensive care units from four institutions, and 120 patients are required to validate the investigators hypothesis. New technologies for the rapid diagnosis of severe infections are investigated in an ancillary study.

ELIGIBILITY:
Inclusion Criteria:

* Major Subject;
* Subject having a sepsis engraves(burns) defined according to the following criteria during the initiation of the probability antibiotic treatment:
* Criteria of SIRS [ 14 ],
* And a suspected infection,
* And a failure of organ: low blood pressure, respiratory failure, coma, hepatic insufficiency, renal insufficiency, thrombopénia, spontaneous extension of the TCA,
* Subject for which an antibiotic treatment was begun within 6 hours following the diagnosis of sepsis engraves(burns);
* Subject for which a taking with microbiological aim was made within 48 hours following the diagnosis of sepsis

Exclusion Criteria:

* Minor Subject, pregnant or breast-feeding woman;
* Neutropénia (PN < 1000 / mm3);
* Absence of identification of a microorganism in the microbiological examinations;
* Absence of Social Security;
* Subject deprived of freedom or under guardianship;
* Subject for which the lit(enlightened) consent is not collected(taken in) (itself and/or reliable person).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
the length of stay | 24 months
  he deadline in days sold enters the diagnosis of sepsis engrave or toxic shock and the exit of resuscitation.

SECONDARY OUTCOMES:
Mortality in resuscitation | 24 months
  The arisen of the death during the initial phase of stay in resuscitation
Lasted treatment antibiotic | 24 MONTHS
  Deadline in days between the beginning of the initiation of the treatment(processing) antibiotic and the 1st day when the subject is not any more handled by antibiotic
Lasted mechanical ventilation(breakdown) | 24 months
  Deadline in days sold between the implementation and the stop(ruling) of the mechanical ventilation(breakdown)
Lasted administration of catécholamines | 24 months
  The number of days without catécholamines during the stay in resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France